CLINICAL TRIAL: NCT01382615
Title: Evaluation of Immune Parameters and Function in Multiple Myeloma Patients and Healthy Individuals' Blood and Marrow Samples
Brief Title: Protocol to Obtain Blood and Bone Marrow Samples for Myeloma Research
Status: Terminated | Type: Observational
Why Stopped: Unable to fill cohort
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Director, Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Other Study IDs: D1029
Record Dates: First submitted 2010-04-12; First posted 2011-06-27 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15mL of peripheral blood 10mL of bone marrow aspirate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers who have agreed to have a bone marrow and/or blood harvest as part of a donation to a transplant recipient.
- Patients with multiple myeloma: Patients undergoing routine blood draw and bone marrow aspirates as part of their ongoing follow-up care for myeloma at the Norris Cotton Cancer Center of DHMC.

SUMMARY:
The purpose of this study is to collect a blood or bone marrow sample from patients with multiple myeloma and from volunteers without myeloma.

DETAILED DESCRIPTION:
The blood and bone marrow samples will be used in the laboratory to perform focused studies on multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Participant population is multiple myeloma patients over the age of 18 who are undergoing a scheduled bone marrow collection and/or blood drawing procedure as part of their routine treatment or follow up, and healthy volunteers over the age of 18 who have agreed to have a bone marrow and/or blood harvest as part of a donation to a transplant recipient.

Exclusion Criteria:

* Patients, who in the opinion of their physician, would be adversely affected by removal of an extra15ml of blood and /or an extra 10ml of bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at Dartmouth-Hitchcock Medical Center's Norris Cotton Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cancer cell response to molecular testing of killing cell parts. | 2 Years
  This myeloma specific killing may help identify mechanisms, in vitro, of killing myeloma cells for the future use in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States